CLINICAL TRIAL: NCT03053596
Title: LifePearl Anthracyclin Registry in Selective Chemo-Embolization of Patients With Unresectable Hepacellular Carcinoma
Brief Title: LifePearl Anthracyclin Registry in Selective Chemo-Embolization of Patients With Unresectable HCC (PARIS Registry)
Status: Completed | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T127E2
Record Dates: First submitted 2016-10-14; First posted 2017-02-15 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; LifePearl
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DEB-TACE using anthracyclin loaded LifePearl™ — The main purpose of this registry is to assess liver toxicity, treatment efficacy, and safety of DEB-TACE using anthracyclin loaded LifePearl™ for treatment of patients with unresectable hepatocellular carcinoma allocated to TACE treatment at multidisciplinary tumor board.

SUMMARY:
The main purpose of this registry is to assess liver toxicity, treatment efficacy, and safety of DEB-TACE using anthracyclin loaded LifePearls for treatment of patients with unresectable hepatocellular carcinoma allocated to TACE treatment.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common type of cancer in men and the eight in women and is the third most common cause of death from cancer worldwide. The overall incidence of HCC remains high in developing countries and is steadily rising in most industrialized countries.

Available treatment options depend on the size, number, and location of tumors; degree of cirrhosis, if present; and comorbidities; overall performance status; patency of portal vein; and presence of metastatic disease. They include surgical (liver resection, liver transplantation), medical (e.g. sorafenib…), ablative (ethanol ablation, radiofrequency ablation, cryoablation) and intra-arterial (chemoembolization, radioembolization) modalities.

Trans Arterial Chemo-Embolization (TACE) with various drugs (anthracyclines being among the most commonly used ones) has been an important therapeutic option for treatment of patients with intermediate stage HCC according to BCLC/EORTC guidelines (REF). In order to maximize therapeutic efficacy of TACE, chemotherapy loadable beads were developed allowing to lower systemic toxicity of chemotherapy, to deliver high and sustained chemotherapy concentration to the tumor, and to prolong delivery of drug and embolization to the tumor.

The purpose of this registry is to evaluate liver and systemic toxicity, treatment efficacy, and safety of Drug Elutable Beads -TACE using anthracyclin loaded Life-Pearls -TACE for unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients, more than 18 years old, with unresectable hepatocellular carcinoma eligible for treatment with anthracyclin loaded LifePearls, allocated to TACE treatment at multidisciplinary tumor board and who agree to data collection in the registry by signing informed consent form.

Exclusion Criteria:

* This is an observational registry and there are no exclusion criteria apart from patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable hepatocellular carcinoma allocated to TACE treatment at multidisciplinary tumor board.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-11; Primary Completion 2019-04-01 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Liver toxicity assessment based on routine CT scans | 12 months

SECONDARY OUTCOMES:
Liver toxicity assessment based on routine blood tests: liver enzymes, phosphatase alkaline, GGT, CBC, bilirubin, albumin. Number of participants with changes in liver function related to TACE treatment. | 12 months
Treatment efficacy based on response rate assessed by mRECIST criteria | 3 months after final TACE
Treatment efficacy based on response rate assessed by RECIST 1.1 criteria | 3 months after final TACE
Safety based on recorded SAE assessed by CTCAE v4.03 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry de Baere, MD, Principal Investigator — Institut Gustave Roussy, France
Locations (7):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - Hôpital Erasme, Brussels
- France (5):
  - Hôpital Beaujon, Clinchamp
  - CHRU Lille, Lille
  - Hôpital Universitaire Saint-Eloi, Montpellier
  - Hôpital L'Archet II, Nice
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Baere T, Guiu B, Ronot M, Chevallier P, Sergent G, Tancredi I, Tselikas L, Dioguardi Burgio M, Raynaud L, Deschamps F, Verset G. Real Life Prospective Evaluation of New Drug-Eluting Platform for Chemoembolization of Patients with Hepatocellular Carcinoma: PARIS Registry. Cancers (Basel). 2020 Nov 17;12(11):3405. doi: 10.3390/cancers12113405. PMID 33212917